CLINICAL TRIAL: NCT00283985
Title: Phase II Study of an Association of L-asparaginase-Methotrexate-Dexamethasone for Relapsing and/or Refractory Nasal and Nasal-type NK-T-cell Lymphoma
Brief Title: Association of L-asparaginase-Methotrexate-Dexamethasone for Nasal and Nasal-type Natural Killer (NK)-T-cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I05009
Record Dates: First submitted 2006-01-30; First posted 2006-01-31 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: NK/T-cell lymphoma; Lymphoma; L-asparaginase; Nasal NK-cell lymphoma; Nasal-type NK-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Extranodal NK-T-Cell; Lymphoma | interventions — Asparaginase; Methotrexate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Kidrolase — 6000 u/ m2 IM at J2, J4 and J6 and J8. 3 to 6 cycles.
Drug: Methotrexate — 3 gr/m2 at J1
Drug: Dexamethasone — 40 mg/ per os at J1, J2 and J4.
Drug: Erwinase — In case of allergy to Kidrolase
  20000 u/m2 en IM at J2, J4, J6 et J8. 3 to 6 cycles

SUMMARY:
Nasal/nasal type NK-T-cell lymphoma is a rare and severe type of non-Hodgkin's lymphoma (NHL) more frequent in Asia than in western countries. When localised, radiotherapy seems to be the best treatment. When radiotherapy cannot be used because of dissemination or relapse, chemotherapy protocols used for other types of NHL give poor results and survival is poor. Recently papers from China and Japan reported the efficacy of a drug: l-asparaginase, usually used to treat acute lymphoblastic leukemia. In vitro a selective apoptosis of NK-cell tumours by l-asparaginase was shown on tumour cell lines and samples.

The investigators propose a phase II protocol for patients with refractory or relapsing nasal/nasal type NK-T-cell lymphoma using a regimen combining l-asparaginase, methotrexate and dexamethasone. Biological studies will be conducted trying to find factors which could predict responses to this chemotherapy.

Since january 2009, the study concerns all patients with nasal/nasal type NK-T-cell lymphoma who have not received asparaginase before.

DETAILED DESCRIPTION:
Primary Objective:

* Determine the overall and complete response rate

Secondary Objectives:

* To evaluate survival without progression
* To evaluate total survival.
* To evaluate the tolerance and the side effects of the treatment.
* To evaluate the duration and the mode of hospitalization of the patients treated by this therapeutic association.
* To constitute a bank of biological samples - serum, tumoral, ADN, ARN to allow prognostic studies implying virus EBV, p53, CD94, C-kit and asparagine synthetase gene in order to better understand the mechanisms of the cancerogenesis of this variety of cytotoxic LNH and to identify the predictive factors of response to the asparaginase.

Sampling:

For each patient included in the protocol, the following sampling will be carried out with the diagnosis:

* Biopsy,
* Medullary biopsy
* Medullary aspiration
* blood: 3 tubes of 7 ml on EDTA and 3 tubs of 7 ml with heparin

Treatment:

All the patients included will receive three cures separated by 3 weeks (J1, J22, J43):

* J1: Methotrexate 3 gr/m2
* J2, J4, J6 and J8: Kidrolase® 6000 u/m2
* J1 with J4: Dexamethasone 40 mg (20 mg if age > 70 years)

ELIGIBILITY:
Inclusion Criteria:

Patients with relapsing/refractory T-NK/NK lymphoma:

* Ages 18 years and above
* Patients must have a diagnosis of NK-cell (or T-NK) non-Hodgkin's lymphoma, nasal or nasal-type.
* Stage I, II, III, or IV disease
* Creatinine less than 3 x upper limit of normal (ULN)
* Able to give informed consent
* No prior treatment with asparaginase

Patients with T-NK/NK lymphoma (de novo patients ):

* Ages 18 years and above
* Patients must have a diagnosis of NK-cell (or T-NK) non-Hodgkin's lymphoma, nasal or nasal-type.
* Stage I, II, III, or IV disease
* Creatinine less than 3 x upper limit of normal (ULN)
* Able to give informed consent
* no prior chemotherapy or radiotherapy

Exclusion Criteria:

* Patients who are pregnant or nursing
* Any factor which might limit the patient's ability to provide informed consent
* Liver insufficiency
* Evolutive thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of chemotherapy | 3 month, 6 month, 9 month, 12 month, 18 month, 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud JACCARD, MD, Principal Investigator — University Hospital, Limoges
Locations (25):
- France (25):
  - Département Maladies du Sang, Angers
  - CH Annecy, Annecy
  - Service de Radiothérapie, Polyclinique Bordeaux Nord, Bordeaux
  - CHU Bordeaux, Bordeaux
  - Service d'Hématologie Clinique - Hôpital Henri Mondor, Créteil
  - Service d'Hématologie Clinique, CHU Dijon, Dijon
  - Service d'Hématologie, Évry
  - CHU Grenoble-Hématologie Clinique, Grenoble
  - CHU Lille - Maladies du Sang, Lille
  - Service d'Hématologie et de Thérapie Cellulaire - CHU Limoges, Limoges
  - CH Lorient, Lorient
  - CHU Lyon - Hématologie Clinique, Lyon
  - Département d'Oncologie - Institut Paoli Calmettes, Marseille
  - CHU Montpellier, Montpellier
  - Hématologie Adulte, Hôpital Necker, Paris
  - Département d'Immuno-Hématologie, Hôpital Saint-Louis, Paris
  - CH Lariboisière, Paris
  - Hôpital St Antoine, Paris
  - Service d'Hématologie Clinique, Groupe Hospitalier Necker, Paris
  - Service d'Hématologie Clinique, Groupe Hospitalier Pitié-Salpétrière, Paris
  - Service d'Immunologie Clinique 2, Hôpital Saint Louis, Paris
  - Service d'Hématologie Clinique, CHU de Reims, Reims
  - Centre Henri Becquerel-Rouen, Rouen
  - Département Hématologie Clinique, Saint-Etienne
  - CHU Toulouse, Toulouse

REFERENCES:
- [Derived] Jaccard A, Gachard N, Marin B, Rogez S, Audrain M, Suarez F, Tilly H, Morschhauser F, Thieblemont C, Ysebaert L, Devidas A, Petit B, de Leval L, Gaulard P, Feuillard J, Bordessoule D, Hermine O; GELA and GOELAMS Intergroup. Efficacy of L-asparaginase with methotrexate and dexamethasone (AspaMetDex regimen) in patients with refractory or relapsing extranodal NK/T-cell lymphoma, a phase 2 study. Blood. 2011 Feb 10;117(6):1834-9. doi: 10.1182/blood-2010-09-307454. Epub 2010 Dec 1. PMID 21123825